CLINICAL TRIAL: NCT03757182
Title: Digitally-Captured Step Counts for Evaluating Performance Status in Advanced Cancer Patients: A Single Cohort, Prospective Trial
Brief Title: Digitally-Captured Step Counts for Evaluating Performance Status in Advanced Cancer Patients
Acronym: DigiSTEPS
Status: Active, not recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Gillian Gresham, Principal Investigator, Cedars-Sinai Medical Center
Other Study IDs: IIT2018-19-GRESH-DIGISTEP
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Cancer; Cancer, Metastatic; Neoplasms
Keywords: Wearable device; Fitness tracker; Wearable activity monitor; Biosensor; Performance Status; Activity Monitoring
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Fitness Trackers; Wearable Electronic Devices; Biosensing Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wearable activity monitor: Continuous activity monitoring with Fitbit Charge HR from baseline to up to 1 year from end-of-study.
  Interventions: Other: Wearable activity monitor

INTERVENTIONS:
Other: Wearable activity monitor — Continuous monitoring of physical activity including step counts, sleep, heart rate, with consumer-based wearable activity monitor (Fitbit Charge HR)
  Other Names: Fitness tracker; Wearable device; Biosensor

SUMMARY:
The purpose of this study is to examine the relationships between objectively measured physical activity and provider-assessed and patient-reported functional outcomes in patients with advanced cancer. Findings from this study will help us better understand how change in daily physical activity, as measured using the wearable activity monitor, is related to change in a patient's functional status and clinical condition.

DETAILED DESCRIPTION:
Patients diagnosed with stage 3/ 4 cancer will be enrolled. After providing informed consent, patients will be asked to wear a FitBit Charge HR continuously for 8 weeks with the option to continue wearing the monitor for up to a year after end-of-study. Baseline assessments include a physical exam, medical history, and frailty assessment. The attending oncologist will rate the patient's performance status (ECOG PS) at baseline and 8-weeks follow-up. Patient-reported outcomes (self-reported physical function, fatigue, sleep, emotional distress) will be assessed weekly using NIH PROMIS from baseline up to 8 weeks from end-of-study. They will also be collected at 1 year follow-up. Wearable activity monitor data will be summarized each week for 8 weeks, and then again at 1 year follow-up. Physical activity data (number of steps, stairs climbed, active minutes, heart rate, and sleep duration) will be collected and analyzed at end-of-study (up to 1 year from end-of-study). Overall survival will also be assessed up to 1 year from end-of-study. Absolute change in physical activity levels will be correlated with change in performance status and occurrence of AEs and death to better understand the role of remote activity monitoring in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced (stage 3 or 4) cancer of any type
* Ambulatory (use of walking aids, such as cane and rollator, is acceptable)
* Access to a device that has the capability to sync to the Fitbit
* Expected to have standard of care oncology appointments at least once every 8 weeks (+/-7 days).
* Have an understanding, ability, and willingness to fully comply with study procedures and restrictions
* English or Spanish speaking
* Ability to consent
* Informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Allergy to surgical steel or elastomer/rubber
* Using a pacemaker, implantable cardiac defibrillator, neurostimulator, implantable hearing aids, cochlear implants, or other electronic medical equipment. However, removable hearing aids are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage 3/4 advanced cancer patients being seen for treatment at Cedars-Sinai Medical Center.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Absolute change in average step counts at 8 weeks from baseline | 8 weeks
  Change will be calculated based on difference in average weekly step count at baseline from the average weekly step count at end-of-study visit
Absolute change in provider-assessed ECOG Performance Status at 8 weeks from baseline | 8 weeks
  Change in performance status will be calculated based on difference in provider-assessed Eastern Cooperative Oncology Group (ECOG) performance status at end-of-study visit and baseline ECOG. ECOG Performance Status is rated based on a 5-point scale where a score of 0 indicates best performance status and 5 indicates death. Only one rating of ECOG PS by provider is completed at each timepoint.

SECONDARY OUTCOMES:
Absolute change in patient-reported physical function at 8 weeks from baseline | 8 weeks
  Physical function will be assessed using the NIH Patient-Reported Outcomes Measurement Information System (PROMIS) short form, which includes 20 items and a range of 1 (low physical function) to 5 (high physical function). The total score will be calculated and converted into a standardized t-score will be calculated based on a standard cancer population with a mean of 50 and SD of 10.
Patient weekly distress levels up to 8 weeks from baseline | 8 weeks
  Distress will be measured using using NIH Patient-Reported Outcomes Measurement Information System (PROMIS), which includes short forms: emotional distress, sleep quality, pain, and fatigue. Items range from 1 (worse outcome) and 5 (best outcome) where a total score will be calculated and converted into standardized t-scores.
Adherence to wearing the device for the specified study period | 8 weeks
  A patient is considered adherent if they wear the device at least 10 hours per day for at least 4 of 7 days prior to each study timepoint
Change in frailty status from baseline to end-of-study visit (up to 8 weeks from baseline) | 8 weeks
  Score calculated based on total number of frailty characteristics present using Fried's validated Frailty index. Characteristics of frailty include shrinking (weight loss), weakness (grip strength), poor endurance, exhaustion, slowness, and low activity. The minimal score is 0, indicating absence of frailty, and the highest is 5. Frailty index categories include absence of frailty (score of 0), pre-frail or intermediate frail (1-2 criteria) and frail (>3 criteria present).
Occurrence of grade 3 or 4 SOC cancer-related adverse events or chemotoxicities and hospitalizations occurring from baseline up to 12 weeks | up to 12 weeks
  AEs will be rated using CTCAE v5
Overall survival up to 1 year from end-of-study | up to 1 year
  Occurrence of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Gresham, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD available upon request.